CLINICAL TRIAL: NCT06185777
Title: Multi-professional Care Pathway and Network for the Promotion of Needs-oriented, Resident-oriented Exercise Therapy for Oncological Patients
Acronym: MOVE-ONKO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Joachim Wiskemann, Prof. Dr. Joachim Wiskemann, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S-571/2023
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Exercise; Implementation
Keywords: Cancer; Cancer treatment; Exercise; Physical Activity; Counseling; Cancer Care; Implementation; Nursing
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise oncology counseling and referal (Experimental): Identification & brief consultation Screening: Needs assessment for exercise therapy Information / educational talk Consultation with the patient Risk assessment (with physician clearance) Consultation Referral to exercise therapy
  Interventions: Behavioral: Exercise oncology counseling and referal

INTERVENTIONS:
Behavioral: Exercise oncology counseling and referal — Identification & brief consultation Screening: Needs assessment for exercise therapy Information / educational talk Consultation with the patient Risk assessment (with physician clearance) Consultation Referral to exercise therapy

SUMMARY:
MOVE-ONKO is developing and implementing a guideline-based, multi-professional care pathway for the promotion and therapy of exercise for cancer patients. This pathway intended to serve as an interface between oncological care and existing or developing exercise therapy services in the local area of the participating hospitals. Needs- and side-effect-oriented care pathways are intended to give as many patients as possible access to quality-assured exercise therapy services close to home and thus to the supportive potential of exercise. The new care pathway will be develop in year 1 (phase 1) and will be established at 7 Comprehensive Cancer Centers (CCCs) in 3 model regions Heidelberg-Frankfurt-Mainz, Dresden-Berlin and Freiburg-Tübingen (phase 2) in Germany, as well as adapted accordingly in organ cancer centers and with established oncological care providers (phase 3 - Outreach). The aim is to ensure that exercise promotion and therapy can be integrated into standard care as comprehensively and sustainably as possible.

The implementation project will be evaluated according to the achievement of implementation and intervention goals. The implementation goals are utilization (reach) and actual implementation. Factors for successful implementation will be identified and incorporated into the procedure in phase 3 (outreach). Intervention goals are mapped at provider and patient level in both phases. They include improving physical functioning, increasing physical activity behavior, improving exercise-related health literacy, increasing motivation to exercise and increasing patient participation. For this purpose, patients with a cancer disease undergoing acute therapy aged 18 and over who are cared for in participating centers are surveyed four times over a period of 24 weeks using standardized questionnaires (baseline (t0) before the intervention, follow-up after 4 (t1), 12 (t2) and 24 (t3) weeks). In addition, the participating managers and service providers of the centers in phase 2 (implementation phase) and phase 3 (outreach phase) will be surveyed using standardized questionnaires and in-depth interviews. The longitudinal evaluation design enables an analysis of the changes in care structures and processes, the success of implementation and the experiences and outcomes of patients

ELIGIBILITY:
Inclusion Criteria (patients):

* cancer patients during chemotherapy, immune therapy or radiotherapy
* having symptoms/side effects that can be effectively treated by exercise (e.g. fatigue) and/or are interested in exercise oncology counseling

Inclusion Criteria (care providers)

- involved in the implementation process

Exclusion Criteria (both):

- Insufficient German language skills

Exclusion Criteria (care providers only):

- Duration employed <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to week 12 in physical function measured by the EORTC QLQ-C30 | baseline till week 12 (& 12 week follow up)
  Physical Function will be assessed within the validated 30-item self-assessment questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30, version 3.0). It comprises five multi-item functional scales (physical, role, emotional, cognitive, and social function), three multi-item symptom scales (fatigue, pain, nausea/vomiting), and six single items assessing further symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea) and financial difficulties. Scores range from 0 to 100. A higher score for the functional scales and global health status denote a better level of functioning, whereas a high score for symptom/single-item scale indicate a higher level of symptomatology/problems. Change = (Week 12 Score - Baseline Score)

SECONDARY OUTCOMES:
Change from baseline to week 12 in physical activity measured by the Godin-Shephard Leisure Time Physical Activity Questionnaire | baseline till week 12 (& 12 week follow up)
  The Godin Leisure-Time Exercise Questionnaire assesses self-reported physical activity (PA) among adults in minutes per week (3 intensity categories: low, moderate, vigorous)
Change from baseline to week 12 in physical activity-related health competence | baseline till week 12 (& 12 week follow up)
  The questionnaire is based on the physical activity-related health competence (PAHCO) model by Sudeck and Pfeifer et al. 2016 and supposed to assess specific facets of the PAHCO, specifically addressing an individual's aptitude to effectively utilize physical activity to optimize their overall health. The questionnaire consists of 13 items comprised of three latent factors: PA-specific mood regulation (MR) (four items), control competence for physical training (CC) (six items) and PA specific self-control (SC) (three items)
Change from baseline to week 12 in social support | baseline till week 12 (& 12 week follow up)
  The Modified Medical Outcomes Study Social Support Survey (mMOS-SS) is an 8-item self-reported measure of individual experience of social support, with two subscale measures of emotional support, and instrumental support. Items ask respondents about having someone to help with physical needs, and emotional assistance. The mMOS-SS is an abbreviated adaptation of the original 19-item
Change from baseline to week 12 in patient activation | baseline till week 12 (& 12 week follow up)
  PAM is a validated questionnaire designed to measure the knowledge, skills and confidence that a person has to manage their own wellbeing (patient activation).
Patients' Experiences Across Health Care Sectors at week 12 | week 12
  The Patients' Experiences Across Health Care Sectors (PEACS) questionnaire is a validated questionnaire to asses patient orientation in a fragmented health-care system
Patients' Shared Decision-Making experience at week 12 | week 12
  The 9-item Shared Decision Making Questionnaire was developed in a theory-driven manner and measures the extent to which patients are involved in the process of decision-making from the perspective of the patient (patient version SDM-Q-9) and from the perspective of the physician (physician version SDM-Q-Doc). The measure was developed for use in research and clinical practice.
Reasons for discontinuing physical/exercise therapy at week 12 and follow-up | week 12 (& 12 week follow up)
  The Problematic Experiences of Therapy Scale (PETS; Kirby, Donovan-Hall, & Yardley, 2014) is a brief measure that was developed based on clinical experience and research to reflect the most commonly reported reasons for discontinuing physical therapy given by patients undergoing self-managed home-based rehabilitation. he PETS comprises 12 Likert-scaled items divided into four subscales: 1. Symptoms too severe or aggravated by therapy (items 1-3), 2. Uncertainty about how to carry out the treatment (items 4-5), 3. Doubts about treatment efficacy (items 6-8), and 4. Practical problems (items 9-12). Each item asks respondents the extent to which they agree that they have been prevented from carrying out an intervention by plausible reasons.
Cancer Patients Information Needs at week 12 and follow-up | week 12 (& 12 week follow up)
  Cancer Patients Information Needs" scale is a validated 17-item questionnaire (Mesters et al. 2001) assessing the various needs of cancer patients during and after cancer treatment
Qualitative interviews and quantitative assessments with the RE-AIM framework to assess quality of pathway structure, processes and efficacy | baseline till week 12 (& 12 week follow up)
  Various measures specific to the implemented intervention

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (7):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Nationales Centrum für Tumorerkrankungen, Heidelberg, Baden-Wurttemberg
  - Medizinische Klinik der Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitäres Centrum für Tumorekrankungen Frankfurt, Frankfurt am Main, Hesse
  - Universitäres Centrum für Tumorerkrankungen Mainz, Mainz, Rhineland-Palatinate
  - Nationales Centrum für Tumorerkrankungen Dresden (NCT/UCC), Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blutgen S, Tigges AL, Zinkevich A, Krug K, Wensing M, Graf K, Wiskemann J, Ansmann L; MOVE-ONKO Consortium. 'It only works if we coordinate our work, that's what we need': a relational qualitative network analysis of exercise therapy in oncology care in Germany. BMC Cancer. 2025 Nov 29;25(1):1845. doi: 10.1186/s12885-025-15326-y. PMID 41318435
- [Derived] Blutgen S, Krug K, Graf K, Betz U, Bohm J, Jager E, Krell V, Muller J, Pahl A, Voland A, Weigmann-Fassbender S, Zinkevich A, Wensing M, Ansmann L, Wiskemann J. Implementation and evaluation of a multi-professional care pathway and network for the promotion of needs-oriented, resident-oriented exercise therapy for oncological patients (MOVE-ONKO): protocol of a mixed-methods cohort study. BMC Cancer. 2025 Mar 13;25(1):458. doi: 10.1186/s12885-025-13797-7. PMID 40082847
- See also: Project Website (in German only) — https://move-onko.de/